CLINICAL TRIAL: NCT00739193
Title: A Randomized, Placebo-Controlled, Double-Blind, Double Dummy Trial To Determine The Relative Effect Of Pm101 Versus Placebo And Amiodarone IV On Blood Pressure In Subjects With Stable Congestive Heart Failure
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Prism Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Baxter Healthcare Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 105
Record Dates: First submitted 2008-08-20; First posted 2008-08-21 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Blood Pressure
Keywords: Blood Pressure
MeSH Terms: interventions — Amiodarone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo Control
  Interventions: Drug: amiodarone
- PM101 (Experimental): PM101
  Interventions: Drug: amiodarone
- Amiodarone IV (Active Comparator): Amiodarone IV
  Interventions: Drug: amiodarone

INTERVENTIONS:
Drug: amiodarone

SUMMARY:
The primary objective of this trial is to compare the relative hemodynamic effect of a novel intravenous formulation of amiodarone (PM101), administered as an immediate IV bolus push, with placebo and with the currentlyl available formulation of Amiodarone IV, administered as a 10-minute IV infusion, on systolic arterial pressure.

ELIGIBILITY:
Inclusion Criteria:

* Men and women >18 years of age at Screening, with a diagnosis of stable congestive heart failure
* NYHA Functional Classification of Heart Failure Class II, III, or IV
* Documented left ventricular ejection fraction ≤35% within 6 months before Screening, provided that the assessment was not within 4 weeks of a myocardial infarction
* Outpatient or inpatient
* On stable doses of medications to treat congestive heart failure (eg, beta-blockers, angiotensin-converting enzyme inhibitor/angiotensin-receptor antagonist, diuretic) for at least 7 days before dosing with trial drug
* Have a 12-lead electrocardiogram (ECG) at Screening that shows no clinically significant abnormalities of rate, rhythm, or conduction (such as high-grade atrioventricular block, bifascicular or trifascicular block), that would jeopardize the safety or the ability to accurately measure the arterial pressure of the subject, in the opinion of the investigator
* Able to communicate effectively with the trial personnel
* Able to undergo study related procedures as required by the protocol
* Adequately informed of the nature and risks of the trial and give written informed consent prior to undergoing any trial-related procedures
* Women of childbearing potential must have a negative pregnancy test both at Screening and at check-in to the trial site before receiving trial drug on Day 1 and must be using an effective medically acceptable form of birth control for the duration of the trial (up through the Day 8 follow-up evaluation)

Exclusion Criteria:

* Known hypersensitivity or allergy to amiodarone, Captisol, Amiodarone IV, or any of its excipients
* Known hypersensitivity or allergy to iodine or radio-opaque dyes
* Presence of asthma or other pulmonary disease, thyroid disease (hypo or hyperthyroidism), hepatitis, or other liver disease that would place the subject at increased risk from treatment with amiodarone, in the opinion of the investigator
* Myocardial infarction within the 30 days before Screening
* Functioning pacemaker at Screening or on Day 1
* Amiodarone administration within 7 days before dosing with trial drug
* Cardiogenic shock, marked sinus bradycardia, or second- or third-degree atrioventricular block
* Any disease or condition that might compromise trial evaluations or place the subject at increased risk from treatment with amiodarone, in the opinion of the investigator
* Any clinically significantly abnormal laboratory test at Screening or Day 1 that would place the subject at increased risk from treatment with amiodarone, in the opinion of the investigator
* Women who are pregnant or breastfeeding A-ny subject who has received an investigational drug within 30 days before dosing with trial drug
* Inability to obtain 3 baseline SAP readings with no more than 5 mm Hg difference among these readings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-08; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure | 15 minutes